CLINICAL TRIAL: NCT00639405
Title: Localization of Parathyroid Adenomas Using MRI and SPECT Fusion Software in Patients With Persistent or Recurrent Hyperparathyroidism
Brief Title: Evaluation of MRI and SPECT Fusion Software to Localize Parathyroid Adenomas
Status: Terminated | Type: Observational
Why Stopped: Subject population not available.
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Michele Lisi, MD, SUNY Upstate Medical University
Other Study IDs: SUNYUMU 5260
Record Dates: First submitted 2008-03-12; First posted 2008-03-20 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2008-10

CONDITIONS: Parathyroid Neoplasm; Parathyroid Diseases
Keywords: Parathyroid; MRI; SPECT
MeSH Terms: conditions — Parathyroid Neoplasms; Parathyroid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: subjects who are diagnosed with parathyroid adenomas. There will be 6 subjects who have not had surgery and 25 subjects who have had surgery.

SUMMARY:
The purpose of this study is to design a method to better localize parathyroid adenomas. This study will include approximately 6 patients who have not had surgery and another 25 patients who have already had surgery over the course of one year.

DETAILED DESCRIPTION:
While a successful neck exploration for PHP is primarily dependent on the experience of the surgeon, there are currently several localizing studies available to increase success. Although the necessity of localizing studies pre-operatively for first time neck explorations is still under debate, there is no question of their importance for persistent or recurrent PHP that requires re-operation. Localizing studies in these patients have been clearly shown to reduce operating time, avoid unnecessary dissection, reduce morbidity, and improve success rate.

Several modalities have been employed for localization such as ultrasound (US), computed tomography (CT), and magnetic resonance imaging (MRI). The sensitivity of ultrasound for the preoperative detection of parathyroid adenomas has been reported to be 65-90% (1). There are however, limitations to US. Because of the sonolucent appearance of parathyroid adenomas, it is impossible to distinguish an ectopic cervical parathyroid adenoma from a pathologic lymph node. Furthermore, mediastinal parathyroid adenomas are difficult, if not impossible to visualize due to acoustic shadowing from the sternum and clavicles (2). Also, this method is very operator-dependent. MRI has a slightly higher sensitivity of 62.5-94% while CT has a poor sensitivity of only 40-44% (1).

We are using dual-phase single photon emission tomography (SPECT) imaging with technetium 99m sestamibi and visual thyroid subtraction with technetium 99m as pertechnetate. This method can achieve sensitivities of 68-95% and specificities of 75-100% (1). SPECT imaging is dependent on the differential washout of sestamibi between normal thyroid tissue and abnormal parathyroid tissue. Theoretically, sestamibi will washout of normal thyroid tissue much more quickly than it will from abnormal parathyroid tissue. Therefore, SPECT imaging is usually performed immediately and then at 90 and 180 minutes after sestamibi injection. SPECT imaging, however, has several limitations, not the least of which is its inability to provide discrete anatomic detail.

In addition, we will use a control group of patients who have parathyroid adenomas but who have not yet had surgery to test the efficacy of our fusion software.

Our goal is to acquire MRI and SPECT imaging with fiducial markers and utilize fusion software to create a detailed anatomic map of the neck for more accurate localization of the lesion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 years and over
* subjects who have had a failed parathyroidectomy and now presents with persistent hyperparathyroidism or recurrent hyperparathyroidism
* 6 control patients with parathyroid adenomas who have not yet had surgery will be selected to test the efficacy of the software.

Exclusion Criteria:

* Potential female subjects who are pregnant
* Any potential subject who has an implanted metallic device, stent or staples
* any subject weighing 300lb

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the Health Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Lisi, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States